CLINICAL TRIAL: NCT00315536
Title: Echocardiographic Study of the Haemodynamic Effects of Remifentanil With and Without Glycopyrrolate in Healthy Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006/042
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Urological Surgery
MeSH Terms: interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of remifentanil and glycopyrrolate — 2 mg, intravenius use

SUMMARY:
Study to investigate the influence of remifentanil and glycopyrrolate on cardiac index and blood pressure in children.To differentiate between contractility and the effect of the circulating volume, some of the subjects will receive additional fluid.This will be evaluated using two transthoracic echocardiac exams within the first 30 min of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II children
* 1-6 years
* urological surgery

Exclusion Criteria:

* Cardiac disease
* Diabetes

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Cardiac index | Twice in 16 minutes.
Blood pressure | Twice in 16 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Reyntjens, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be